CLINICAL TRIAL: NCT03762642
Title: Trends of Mastectomy and Breast-Conserving Surgery and Related Factors in Female Breast Cancer Patients Treated at King Abdulaziz University Hospital, Jeddah, Saudi Arabia, 2009-2017
Brief Title: Trends of Mastectomy and Breast-Conserving Surgery in Female Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Zuhoor K. AL-Sharif, Professor, King Abdulaziz University
Other Study IDs: 357-71
Record Dates: First submitted 2018-11-30; First posted 2018-12-04 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Breast Cancer; Breast Neoplasms; Breast Cancer Female
Keywords: Breast Cancer Surgery; Lumpectomy; Surgery Choice; Procedure Choice; Surgical Outcome
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy; Mastectomy, Segmental

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mastectomy
  Interventions: Procedure: Mastectomy
- Breast-Conserving Surgery
  Interventions: Procedure: Breast-Conserving Surgery

INTERVENTIONS:
Procedure: Mastectomy — Removal of the whole breast
  Groups: Mastectomy
Procedure: Breast-Conserving Surgery — Removal of the cancerous tissue only
  Other Names: Lumpectomy
  Groups: Breast-Conserving Surgery

SUMMARY:
Breast cancer is the most common cancer in women across the world, accounting for 25.2% of cancer cases among females and 14.7% of cancer-related deaths among females worldwide. The survival rates are markedly lower in the developing countries compared to developed countries, as well as the age at diagnosis. Core management of breast cancer includes surgical removal of the tumor either by breast-conserving surgery (BCS) or mastectomy (removal of the whole breast). Choosing between these two procedures may be influenced by factors that have yet to be studied in Saudi Arabia. The investigators aimed to determine the prevalence of BCS and mastectomy and the factors that may influence the choice of procedure. This retrospective study was carried out by reviewing the records of female breast cancer patients who underwent BCS or mastectomy at King Abdulaziz University Hospital between 2009 to June 2017, excluding those with metastasis (distant spread of the cancer) or recurrence. Using frequencies for the rate, and multivariate tests, the investigators analyzed different demographic, clinicopathological, and radiological factors to detect correlations with procedure choice.

ELIGIBILITY:
Inclusion Criteria:

* Female, diagnosed with breast cancer, underwent surgery on the breast tumor in King Abdulaziz University Hospital

Exclusion Criteria:

* Patients with metastatic breast cancer or recurrence of the cancer before the surgery

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Female breast cancer patients who underwent surgery for breast cancer in King Abdulaziz University hospital between 2009 and June 2017 excluding those who had metastasis or recurrence before the surgery
Sampling Method: Non-Probability Sample
Enrollment: 335 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2018-08-02 (Actual)

PRIMARY OUTCOMES:
Prevalence of each of mastectomy and breast-conserving surgery | 2009-2017
  The percentage of of patients who underwent each surgery

SECONDARY OUTCOMES:
The relationship between the choice of procedure and the patients' age (in years) | 2009-2017
  Statistical analysis using independent sample T-test and binary logistic regression
The relationship between the choice of procedure and the use of preoperative chemotherapy (also called "neoadjuvant chemotherapy") | 2009-2017
  Statistical analysis using Chi-square test and binary logistic regression
The relationship between the choice of procedure and the tumor's laterality (right versus left breast cancer) | 2009-2017
  Statistical analysis using Chi-square test and binary logistic regression
The relationship between the choice of procedure and the tumor's focality (whether it is composed of more than one mass) | 2009-2017
  Statistical analysis using Chi-square test and binary logistic regression
The relationship between the choice of procedure and the tumor's centricity (whether it involves more than one quadrant of the breast) | 2009-2017
  Statistical analysis using Chi-square test and binary logistic regression
The relationship between the choice of procedure and the tumor's size (in centimeters) | 2009-2017
  Statistical analysis using independent sample T-test and binary logistic regression
The relationship between the choice of procedure and the tumor's stage (using the 7th "American Joint Committee on Cancer"'s staging guidelines) | 2009-2017
  Statistical analysis using Chi-square test and binary logistic regression
The relationship between the choice of procedure and the tumor's histological grade (using the Nottingham Histologic Score system) | 2009-2017
  Statistical analysis using Chi-square test and binary logistic regression
The relationship between the choice of procedure and the tumor's receptor status (whether it is positive for estrogen, progesterone, and/or human epidermal growth factor receptor 2) | 2009-2017
  Statistical analysis using Chi-square test and binary logistic regression
The relationship between the choice of procedure and having preoperative magnetic resonance imaging of the breast and its findings | 2009-2017
  Statistical analysis using Chi-square test and binary logistic regression

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Jeddah, Mecca Region, Saudi Arabia